CLINICAL TRIAL: NCT04371731
Title: A Single-centre Research Study to Evaluate the Impact of a Novel Care Pathway for Patients Diagnosed With Heart Failure (HF) Within Chiltern CCG, Supported by an Integrated Clinical Patient Record. Assessment of Patient Outcomes Following Implementation of Care4Today® Heart Failure Platform.
Brief Title: A Single-centre Research Study to Evaluate the Care4Today® Heart Failure Platform.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buckinghamshire Healthcare NHS Trust (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RXQ682
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Intervention Model Description: Two arms, one using the platform to help manage their heart failure and one standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental): Active cohort will use the Care4today platform to help manage their heart failure
  Interventions: Other: Care4todayheart failure platform
- Control arm (No Intervention): Control arm will contain standard of care heart failure treatment

INTERVENTIONS:
Other: Care4todayheart failure platform — Platform allowing patients to enter information about their health at home, namely weight and BP and medications
  Arms: Active Arm

SUMMARY:
A research study to evaluate the impact of a novel care pathway for patients diagnosed with Heart Failure within Chiltern CCG, supported by an integrated clinical patient record. Assessment of patient outcomes following implementation of Care4Today(R) Heart Failure Platform.

DETAILED DESCRIPTION:
This is an exploratory study to evaluate the impact of the novel Care4Today HF platform on a set of outcomes including hospital admission rate (primary diagnosis), 30 days post discharge readmission rate, length of hospital stay for patients with HF (primary and secondary diagnosis), patient quality of life, and patient clinical metrics. The study design includes comparison of two parallel cohorts: one where patients will be managed via the Care4Today HF platform (active cohort) and a second, where patients will be managed as per existing standards of care (control cohort).

Evaluation phase:

The evaluation phase will be set up to assess the potential benefits of the Care4Today HF platform. This will be implemented across 10 GP practices who will be part of the active cohort, within the Chiltern CCG region. The outcomes for these patients will be compared with the outcomes of patients in the control cohort over a one year period.

Patients pathway (for the active cohort):

Once the diagnosis of HF is confirmed, a HF specialist project nurse will register the patient on the Care4Today platform and provide the patient with instructions on how to use the patient portal, where patients can input various clinical measures, communicate with HCPs and track their condition. Complex patients, and/or patients that are deteriorating are referred to the community HF specialist nurse team where they will be monitored and managed.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older with the primary diagnosis of heart failure
* Must have moderate to severe LVSD (ejection fraction <= 40%) confirmed by an echocardiogram and/or other cardiac imaging

Exclusion Criteria:

* Patients with right heart failure as a consequence of respiratory disease
* Patients with Heart Failure with preserved Ejection Fraction
* Patients with significant learning disability, or severe mental health conditions
* Patients with metabolic heart disease e.g. amyloid
* Patients with severe non-operable valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Hospital admissions | 12 months
  number of hospital admissions

SECONDARY OUTCOMES:
mean number of heart failure readmissions within 30 days of discharge | 30 days of discharge
  mean number of heart failure readmissions within 30 days of discharge
all cause readmissions | 12 months
  mean number of all cause readmissions
length of stay | 12 months
  o Mean, median (SD) days of length of stay (for admissions with a primary and secondary diagnosis of HF)
weight change | 12 months
  Mean (SD) change in weight
Blood pressure | 12 months
  o Proportion of patients achieving target for blood pressure (140/90mmHg or 130/80mmHg for patients with diabetes) at the end of the study
Hospital Anxiety and Depression Scale score | 12 months
  Mean change in Hospital Anxiety and Depression Scale (HADS) at the start and after 1 year the end of the study. Score on scale of 0-21, 0-7 = normal, 8-10 borderline, 11-21 abnormal. Higher score = worse outcome
QOL | 12 months
  o Mean change in Quality of Life assessed by Minnesota Living with Heart Failure Questionnaire and EQ5D or EQVAS

IPD SHARING:
Plan to Share IPD: No